CLINICAL TRIAL: NCT00623246
Title: Motivating Adherence to CPAP in Obstructive Sleep Apnea
Brief Title: Evaluating Behavioral Treatments to Improve Adherence to Continuous Positive Airway Pressure (CPAP) Therapy in People With Obstructive Sleep Apnea (The BREATHE Study)
Acronym: BREATHE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Jewish Health (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Center for Research Resources (NCRR) (NIH); The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 560; R01HL067209 (NIH); 2R01HL067209 (NIH)
Record Dates: First submitted 2008-01-07; First posted 2008-02-25 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Sleep Apnea, Obstructive; Continuous Positive Airway Pressure
Keywords: Obstructive Sleep Apnea; OSA; Adherence; CPAP; Cognition
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Participants will receive motivational enhancement therapy (MET) for 12 weeks.
  Interventions: Behavioral: MET
- 2 (Active Comparator): Participants will receive educational therapy (ED) for 12 weeks.
  Interventions: Behavioral: ED
- 3 (No Intervention): Participants will receive standard clinical care.

INTERVENTIONS:
Behavioral: MET — MET will involve motivational counseling sessions and phone calls, with a focus on building self-efficacy and providing personalized feedback on health and adherence patterns based on CPAP adherence monitoring.
  Arms: 1
Behavioral: ED — ED will involve sessions and phone calls that include educational information, problem-solving, and adherence feedback from study staff.
  Arms: 2

SUMMARY:
Obstructive sleep apnea (OSA) is a serious sleep disorder in which a person repeatedly stops breathing or experiences shallow breathing for short periods of time during sleep. The most common treatment for OSA is the use of a continuous positive airway pressure (CPAP) machine, but many people have trouble adhering to the treatment schedule. This study will evaluate the effectiveness of two behavioral therapy programs used in combination with CPAP for improving treatment adherence in people with OSA.

DETAILED DESCRIPTION:
OSA is a common sleep disorder that is characterized by a brief collapse and blockage of the upper airway during sleep. This blockage prevents air from flowing properly into the lungs and causes pauses in breathing. Symptoms include loud snoring, choking or gasping during sleep, and abnormal daytime sleepiness. If left untreated, OSA can lead to heart disease, high blood pressure, and stroke. The most common treatment for OSA is CPAP therapy, in which a mask is worn over the nose during sleep and pressurized air flows through the mask to keep the throat open. Unfortunately, CPAP treatment adherence is often poor. Previous research studies showed that people receiving motivational enhancement therapy (MET) or educational therapy (ED) adhered better to CPAP treatment than did people not receiving MET or ED therapy. However, even for people who received MET or ED, adherence usually diminished after 12 months. It appears that patterns of treatment adherence are often set early and people who maintain adherence within the first week of treatment have a greater chance of maintaining long-term adherence. Using enhanced, more intense versions of MET and ED that are delivered when CPAP therapy begins, this study will evaluate the effectiveness of MET and ED at improving CPAP treatment adherence in people with OSA.

This study will enroll people with OSA. Participants will be randomly assigned to a 12-week MET group, a 12-week ED group, or a standard clinical care group, with all treatments beginning at the time participants start CPAP therapy. All participants will attend a baseline study visit to undergo weight and blood pressure measurements; assessments of cognitive functioning, mood, daytime sleepiness, functional outcomes, and attitudes toward therapy; and an optional blood collection. At baseline and Week 1, participants in the MET and ED groups will take part in two 45-minute, face-to-face counseling sessions. During these sessions, participants in the MET group will receive motivational counseling from study staff, and participants in the ED group will receive educational information about OSA from study staff. At Months 1 and 3, participants will receive two phone calls from study staff. The MET group will receive motivational counseling during these calls, with a focus on building self-efficacy and providing personalized feedback on health and adherence patterns. The ED group will receive educational information and feedback on problem-solving and adherence during the calls. Throughout the study, all participants will have their CPAP adherence electronically monitored on a daily basis. Participants who fail to meet the minimum standard of CPAP adherence will receive up to four additional phone calls during the study. At Months 3, 6, and 12, all participants will attend study visits for repeat baseline measurements.

ELIGIBILITY:
Inclusion Criteria:

* OSA confirmed by polysomnography (PSG)
* CPAP is the prescribed form of treatment for OSA
* Judged by sleep physician to respond to CPAP

Exclusion Criteria:

* Apnea/hypoxia index (AHI) less than 15 and no daytime functional symptoms or associated cardiovascular disease
* Diagnosis of another sleep disorder that causes arousals from sleep
* Past treatment for OSA
* Current substance abuse problem
* Diagnosis of a serious medical condition that would interfere with involvement in the study
* History of a major psychiatric disorder, other than depression
* Change in antidepressant medication in the 3 months before study entry

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2007-12; Primary Completion 2012-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Adherence to CPAP | Measured at Months 3, 6, and 12
Cognitive function | Measured at Months 3, 6, and 12
Subjective sleepiness | Measured at Months 3, 6, and 12
Quality of life | Measured at Months 3, 6, and 12

SECONDARY OUTCOMES:
Blood pressure | Measured at Months 3, 6, and 12
Cytokines and inflammatory markers | Measured at Month 3
Attitudes toward CPAP use (transtheoretical model [TTM] and social cognitive theory [SCT] model variables) | Measured at Months 3, 6, and 12

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Aloia, PhD, Principal Investigator — National Jewish Health
Locations (1):
- National Jewish Medical and Research Center, Denver, Colorado, United States